CLINICAL TRIAL: NCT07165470
Title: Pre-Packaged Low-Residue Diet Assisting Bowel Preparation in Patients With Inflammatory Bowel Disease：A National Multicenter Randomized Controlled Clinical Trial
Brief Title: Pre-Packaged Low-Residue Diet Assisting Bowel Preparation in Patients With Inflammatory Bowel Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHEC2025-312
Record Dates: First submitted 2025-09-01; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Colonoscopy: Bowel Preparation; IBD - Inflammatory Bowel Disease
Keywords: bowel preparation; colonoscopy; IBD - Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Powder Group (Experimental): Participants will be provided with 6 sachets of pre-packaged low-residue diet one day prior to colonoscopy, to be consumed as needed in multiple servings during the day.
  Interventions: Dietary Supplement: pre-packaged low-residue diet for bowel preparation
- Standard Low-Residue Diet Group (No Intervention): Participants follow standard low-residue diet guidelines (like ESPEN recommendations) for 24 hours before colonoscopy. This includes rice water, congee, noodles, and steamed eggs, while avoiding fruits/juices, vegetables, nuts, and other high-fiber foods.

INTERVENTIONS:
Dietary Supplement: pre-packaged low-residue diet for bowel preparation — Participants will be provided with 6 sachets of pre-packaged low-residue diet one day prior to colonoscopy
  Arms: Nutrition Powder Group

SUMMARY:
The primary objectives of this study are as follows:

1.To evaluate the efficacy of Maifu Changqing® Complete Nutritional Formula Powder in bowel preparation for colonoscopy among inflammatory bowel disease (IBD) patients;2.To enhance nutritional status and procedural comfort during bowel preparation in the IBD population.

DETAILED DESCRIPTION:
The project workflow comprises three consecutive phases: In the initiation phase, key activities include designing the study protocol, developing a bowel preparation assessment questionnaire, and establishing collaborative multicenter partnerships. During the implementation phase, subjects will be randomized into two arms-the control arm receiving conventional low-residue diet and the intervention arm administered Maifu Changqing® Complete Nutritional Formula Powder-with both regimens initiated 24 hours prior to colonoscopy. Clinical data will be systematically collected while Case Report Forms (CRFs) from all participating centers are centrally aggregated. The conclusion phase focuses on CRF quality control through standardized verification procedures to ensure data integrity, completeness, and objectivity according to Good Clinical Practice (GCP) standards.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adult patients between 18 and 75 years old;
* Diagnosis of IBD according to the 2023 Guidelines for the Diagnosis and Treatment of Inflammatory Bowel Disease;
* Voluntary participation in this clinical trial and provision of signed informed consent.

Exclusion Criteria:

* Patients with acute IBD, severe conditions, combined with major bleeding, suspected toxic megacolon, CD with severe intestinal stricture, gastrointestinal obstruction, or other conditions deemed unsuitable for colonoscopy by the physician;
* Patients with severe cardiac, pulmonary, hepatic, or renal dysfunction;
* History of previous colorectal surgical resection or use of medications that may affect intestinal motility within one week (e.g., antidepressants, sedatives, calcium channel blockers);
* History of stroke, spinal cord injury, or psychiatric disorders that impair compliance with bowel preparation and colonoscopy;
* Allergy to any component of the administered drugs or meal replacements;
* Pregnant or lactating women, and other individuals considered unsuitable for bowel preparation and colonoscopy by the physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bowel preparation adequacy rate | 6 months
  Bowel preparation adequacy rate:Proportion of subjects with a Boston Bowel Preparation Scale (BBPS) score of ≥2 in each segment.The BBPS ranges from 0 to 3 per segment (total score 0-9), with higher scores indicating better bowel cleanliness.

SECONDARY OUTCOMES:
Subject Satisfaction | 6 months
  Subjects' subjective satisfaction with and willingness to repeat the entire bowel preparation process, assessed using a Visual Analogue Scale (VAS).The VAS is a 100-mm horizontal line anchored at "extremely dissatisfied" (0 mm) and "extremely satisfied" (100 mm). Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Bai, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No